CLINICAL TRIAL: NCT03053401
Title: Ultrasound Guided Single Shot Adductor Canal Block (ACB) Versus Single Shot Femoral Nerve Block (FNB) for Postoperative Analgesia After Arthroscopic Anterior Cruciate Ligament (ACL) Reconstruction in Pediatrics
Brief Title: Ultrasound Guided Adductor Canal Versus Femoral Nerve Blocks for Anterior Cruciate Ligament Reconstruction in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Rami Karroum, Staff Anethesiologist,M.D., Akron Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 001126
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Post-operative Pain; Quadriceps Muscle Strength
Keywords: Quadriceps muscle strength; Anterior cruciate ligament reconstruction; Femoral nerve block; Adductor Canal block; Saphenous nerve block in the Adductor Canal; Pediatrics; Postoperative analgesia; Ultrasound guided nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultrasonography; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal block (Active Comparator): Adductor Canal Block performed at mid-thigh level to block the saphenous nerve under guidance of a linear ultrasound transducer probe (General Electric; GE). Performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg ( maximum of 40 mg ).
  Interventions: Procedure: Adductor Canal Block; Device: Ultrasound; Device: Stimuplex A needle; Drug: local anaesthetic injection; Drug: Steroid Drug
- Femoral Nerve block (Active Comparator): Femoral Nerve Block performed under guidance of a linear ultrasound transducer probe (General Electric;GE).Block will be performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg (maximum of 40 mg ).
  Interventions: Procedure: Femoral Nerve Block; Device: Ultrasound; Device: Stimuplex A needle; Drug: local anaesthetic injection; Drug: Steroid Drug

INTERVENTIONS:
Procedure: Adductor Canal Block — Under guidance of a linear ultrasound transducer probe (General Electric; GE). Performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg ( maximum of 40 mg ).
  Arms: Adductor Canal block
Procedure: Femoral Nerve Block — Under guidance of a linear ultrasound transducer probe (General Electric;GE).Block will be performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg (maximum of 40 mg ).
  Arms: Femoral Nerve block
Device: Ultrasound — Use of linear ultrasound transducer probe (General Electric;GE) to guide needle placement for both Adductor Canal Block and Femoral nerve Blocks
Device: Stimuplex A needle — 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany) used to perform both Adductor Canal Block and Femoral nerve Blocks.
Drug: local anaesthetic injection — Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) for either Adductor Canal Block and Femoral nerve Blocks.
Drug: Steroid Drug — Methylprednisolone acetate 1 mg/kg (maximum of 40 mg ) for either Adductor Canal Block and Femoral nerve Blocks.

SUMMARY:
Both Ultrasound guided Adductor Canal Block ( ACB) and Femoral Nerve Block (FNB) has been used to provide postoperative analgesia for knee surgeries. To the investigators' knowledge, no comparison has been made between those blocks in relation to postoperative quadriceps muscle strength, or duration and quality of postoperative analgesia for arthroscopic ACL reconstruction in pediatrics. If ACB provides postoperative analgesia after arthroscopic knee surgery comparable to FNB, it has the potential to improve the postoperative outcome as it will lead to less quadriceps muscle weakness and early mobilization, both of which are very important in the early postoperative period.

DETAILED DESCRIPTION:
Motor preservation with adequate analgesia has become the optimal postoperative goal in orthopedic surgeries, in particular knee surgeries. This enables earlier physical therapy, faster recovery and shorter hospital stays. Both Ultrasound guided ACB and FNB has been used to provide postoperative analgesia for knee surgeries, including anterior cruciate ligament reconstruction . To the investigators' knowledge, no comparison has been made between both blocks in relation to postoperative quadriceps muscle strength as well as duration and quality of postoperative analgesia for arthroscopic ACL reconstruction. ACB predominantly block the sensory component of the femoral nerve without much effect on the motor component. Hence, it can lead to less quadriceps muscle weakness, early postoperative mobilization and decreases the incidence of postoperative fall . With the advent of ultrasonography, the adductor canal can be easily visualized at the mid-thigh level, allowing performance of ACB with a high success rate . In recent years, ACB has been successfully used for postoperative pain control after knee surgery . Anatomical study of adductor canal demonstrated that the adductor canal may serve as a conduit for more than just the saphenous nerve, possibly including the vastus medialis nerve, medial femoral cutaneous nerve, articular branches from the obturator nerve, as well as the medial retinacular nerve . Thus, the sensory change is not limited to the distribution of the saphenous nerve but includes the medial and anterior aspects of the knee from the superior pole of the patella to the proximal tibia.To the investigators Knowledge there has not been a randomized controlled study comparing ACB with FNB after Arthroscopic Anterior Cruciate Ligament (ACL) reconstruction. This prospective, double-blinded, randomized, controlled study will test the hypothesis that ACB would be associated with less quadriceps motor weakness than FNB at 4 hours after block performance . The investigators also hypothesize that ACB will provide analgesia to the anterior knee that is not inferior to FNB and not different in opioids usage at 4 and 24 hours after Peripheral Nerve Block (PNB) performance .

* Hypothesis ACB would be associated with less quadriceps motor weakness than FNB and provide postoperative analgesia comparable to FNB in quality and duration as determined by Numeric Scale (NS) pain scores and opioid use a 4 and 24 hours after PNB.
* Objectives

To compare FNB and ACB regarding:

1. Quadriceps muscle strength at 4 hours after PNB performance.
2. Pain scores at anterior knee at 4 hours and 24 hours after PNB as assessed by Numeric Scale (NS) pain scoring system. Also pain site other than the anterior knee will be recorded and specified (posterior knee, calf, leg)
3. Total opioid consumption at 4 and 24 hours after PNB.

   * Study Design:

Randomized, double blinded, single center clinical trial. A total of 52 pediatric patients (ASA 1or 2), aged between 8 to 18 years, for elective ACL reconstruction at Akron Children's Hospital ( ACH ) will be enrolled in the study. Patients will be randomly assigned to one of two groups, A or B. Group A (26 patients) will have ultrasound guided ACB performed at mid-thigh level and group B (26 patients) will have ultrasound guided FNB, with nerve stimulator confirmation with the type of motor response (e.g., quadriceps, patellar) and the minimum current needed to be recorded. Both blocks will be performed under general anesthesia. Both group will have ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml and methylprednisolone acetate 1 mg/kg , maximum of 40 mg ).Both blocks will be performed using a 22-gauge 2-inch Stimuplex A needle; ; B. Braun Medical Inc., Melsungen, Germany).Both blocks will be performed using linear ultrasound transducer, General Electric ( GE). Ultrasound pictures will be obtained to Verify proper local anesthetic placement.Unfortunately, surgeons are not able to determine the type of procedure needed to correct ACL injury, until after knee arthroscopy is performed under general anesthesia. ACL reconstruction using a hamstring graft, which is the surgical procedure used in this study may not always be possible to perform by the surgeon. The surgical alternative of ACL reconstruction , is ACL repair, which seldomely is done by our surgeon. Patient undergoing ACL reconstruction can experience pain in the posterior aspect of the knee, in the distribution of the siatic nerve. This is due to the hamstring graft. In contrast to the anterior knee pain covered by both ACB and FNB, posterior knee pain is controlled with IV/oral analgesic. This is why recording the site of the knee pain is important to determine the PNB success. . Due to the inability to determine beforehand, the type of procedure to be performed, we decided therefore to continue the study procedures and data collection on both ACL reconstruction and ACL repair. The statistical analysis will include only patients that undergo ACL reconstruction. For the other patients that undergo ACL repair , data will be collected but not included in the statistical analysis. The data from these patients may be used as a pilot for future research.

Quadriceps strength of both legs will be assessed by placing the dynamometer on the anterior of the ankle, between the malleoli. Patients will be instructed to extend their legs three times each, with a 30 seconds pause between each attempt as described by Maffiuletti . The assessment will be performed in the pre-operative period and will be repeated postoperatively at 4 hours after PNB. All patients will be observed in the post-operative period by an observer unaware of the technique of analgesia used. Pain will be assessed using the NS. Postoperatively, PCA morphine pumps will be attached to patients. A loading dose of 0.05 mg/kg to a maximum of 5 mg will be administered in the Post Anesthesia Care unit (PACU) as needed, followed by demand interval dosing of 0.015 mg/kg every 10 minutes.as demanded by the patient .Four-hours limits for morphine will be set at 0.35 mg/kg. No continuous infusion and no adjuvant NSAIDs or acetaminophen will be administered. Rescue morphine dosing will be ordered via PCA pump at 0.05 mg/kg ( repeated once as needed) and will be available every two hours as needed by pain assessment ( for a NS ≥ 4 ) or patient request. Diazepam 0.03 mg/kg IV will be available every 4 to6 hours as needed for muscle spasm or anxiety. Patients will be considered ready for discharge from hospital when all the following criteria are met: Child is alert, oriented, stable vital signs, and would tolerate clear liquid, with no nausea or vomiting and good pain control. The evaluation for meeting the discharge criteria will be done after one hour from arrival in PACU and every 30 minutes thereafter till the patient meet all the discharge criteria. After discharge, After discharge, parents will be instructed to give the child oxycodone tablets/elixir 0.1 mg /kg PO q 3 hours as needed for pain. In addition, acetaminophen 10mg/kg q 4 hours PRN up to a maximum of 3 gm and/or ibuprofen 10 mg/kg q 6 hours PRN up to maximum of 2400 mg/24 hours, may be administered for any residual pain. The total dose of oxycodone, ibuprofen and tylenol will be recorded per parents for a total of 24 hours after PNB. Pain scores will be also recorded by parent at rest,24 hours post -block. The data for total opioids use in the first 24 hours after PNB and pain score at 24 hours will be collected from parent by phone call.

* Study Endpoints

  1-Quadriceps muscle strength at 4 after PNB 2- Total morphine/morphine equivalent at 4 and 24 hours after PNB. 3-Pain scores at anterior knee at 4 hours and 24 hours after PNB as assessed by Numeric Scale (NS) pain scoring system. Also pain site other than the anterior knee will be recorded and specified (posterior knee, calf, leg).
* Method for Assigning Subjects to Treatment Regimen Random allocation for one of the two treatments will be achieved using sealed envelope assigned by external third party not involved in the study to ensure allocation concealment.
* Study Monitoring Plan This study will be monitored through a data monitoring committee. The study will be performed over a period of 18-24 months. This study offers minimal risk to the patient. The data monitoring committee will include the PI, at least one of the co-investigators, the principal statistician, and the principal research nurse.

The data monitoring committee will meet when approximately 25%, 50%, 75% and 100% of the primary outcomes are observed. The priority of the data monitoring committee will be to ensure the safety of the participants in the trial and to ensure the integrity of the trial. Also, these meetings will monitor the quality of the collected data to assess for weaknesses and errors. If any weakness and/or errors are identified, feedback will be provided during these meetings .The investigator(s) will allocate adequate time for such monitoring activities. The investigator(s) will also ensure that the monitor or other compliance or quality assurance reviewer is given access to all the above noted study-related documents.

-Summary Statistics: Will be provided for all variables. Examination of continuous data will include normality testing as well as assessment of potential outliers. Statistical testing will be based upon distributional shape, but for purpose of analytical planning and sample size analysis normality of distributions will be assumed.

To examine for potential differences in quadriceps motor strength (QMS) between the two groups (ACB, FNB) quadriceps strength will be assessed at the four hour time point (assuming no evidence in sample of baseline or pre-operative differences). Non-inferiority of ACB to FNB in analgesia provided will be assessed by examination of pain scores. Non-inferiority of ACB compared with FNB is defined as the mean ACB - NRS pain score not higher than the mean FNB - NRS pain score by an amount of 1.6. (Kim, 2014) Pain scores will be individually examined at the 4 hour and 24 hour post - operative time points with appropriate Bonferroni adjusted alpha. In addition, a change in pain score from 4 to 24 hours will be created and evaluated for potential difference between groups.

Total opioid consumption as measured in morphine equivalents will be assessed at the 24 hour post-operative time point to determine whether a difference exists. Opioid consumption will also be examined by creating a change score from 4 to 24 hour consumption and comparing between the groups.

All testing will be completed utilizing SAS 9.4 © software and evaluated at the Type I Error Rate of alpha = 0.05 level for statistical significance unless otherwise noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Age 8 to 18 years
* All research subjects must have an acceptable legally authorized representative capable of giving consent on the subject's behalf.

Exclusion Criteria:

* Those who were unable to use a standard 0-10 NS
* Infection at the site of the block
* Bleeding disorders
* Allergy to the drugs used to perform the block ( ropivacaine , methylprednisolone)
* Those who refused a nerve block or enrollment in the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Karroum, MD, Principal Investigator — Akron Chidren's hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Result] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Result] Atkinson HD, Hamid I, Gupte CM, Russell RC, Handy JM. Postoperative fall after the use of the 3-in-1 femoral nerve block for knee surgery: a report of four cases. J Orthop Surg (Hong Kong). 2008 Dec;16(3):381-4. doi: 10.1177/230949900801600324. PMID 19126912
- [Result] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Result] Manickam B, Perlas A, Duggan E, Brull R, Chan VW, Ramlogan R. Feasibility and efficacy of ultrasound-guided block of the saphenous nerve in the adductor canal. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):578-80. doi: 10.1097/aap.0b013e3181bfbf84. PMID 19916251
- [Result] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Result] Akkaya T, Ersan O, Ozkan D, Sahiner Y, Akin M, Gumus H, Ates Y. Saphenous nerve block is an effective regional technique for post-menisectomy pain. Knee Surg Sports Traumatol Arthrosc. 2008 Sep;16(9):855-8. doi: 10.1007/s00167-008-0572-4. Epub 2008 Jun 24. PMID 18574578
- [Result] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Result] Krombach J, Gray AT. Sonography for saphenous nerve block near the adductor canal. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):369-70. doi: 10.1016/j.rapm.2007.04.006. No abstract available. PMID 17720129
- [Result] Maffiuletti NA. Assessment of hip and knee muscle function in orthopaedic practice and research. J Bone Joint Surg Am. 2010 Jan;92(1):220-9. doi: 10.2106/JBJS.I.00305. PMID 20048117
- [Result] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- [Result] Luo TD, Ashraf A, Dahm DL, Stuart MJ, McIntosh AL. Femoral nerve block is associated with persistent strength deficits at 6 months after anterior cruciate ligament reconstruction in pediatric and adolescent patients. Am J Sports Med. 2015 Feb;43(2):331-6. doi: 10.1177/0363546514559823. Epub 2014 Dec 2. PMID 25466410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be seen in the orthopedic office prior to the scheduled surgery. An informed consent will be provided for review by the authorized legal representative (s). If they agree to participate in the study, they will be requested to sign and date the informed consent.Patient ascent to the study may be also requested if needed.
Period: Overall Study
Arm/Group | Adductor Canal Block | Femoral Nerve Block
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Femoral Nerve Block: Femoral Nerve Block performed under guidance of a linear ultrasound transducer probe (General Electric;GE).Block will be performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg (maximum of 40 mg ).
  .
- Total: Total of all reporting groups
Arm/Group | Adductor Canal Block | Femoral Nerve Block | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 26 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (1.5) | 15.2 (2.0) | 15.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 10 | 11 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Pre-Surgical Quadriceps Muscle Strength [Median (Full Range); unit: kgf] | 18.4 [4.7 to 33.8] | 19.0 [4.9 to 38.3] | 18.8 [4.7 to 38.3]

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength in Kilogram-force (Kgf)
Description: Measuring the quadriceps muscle strength (surgical side) using a dynamometer.Patients were placed supine with a cushion underneath their knee, resulting in a 45-degree angle at the knee. A dynamometer was placed on the anterior of the ankle, between the malleoli. Patients were instructed to extend their legs three times each, with a 30-s pause between each attempt (Lafayette Manual Muscle Test System; Lafayette Instrument Company, Lafayette, IN; and all three dynamometer readings in Kgf unit for each leg were recorded.Kgf is a gravitational metric unit force ,it is equal to the magnitude of the force exerted on one kilogram of mass under standard gravity.
Time Frame: 4 hours following peripheral nerve block performance
Population: 20 of 26 subjects in the femoral nerve block group had recorded quadriceps muscle strength of zero.
Measure: Median (Full Range); unit: Kilogram-force (Kgf)
Groups:
- Adductor Canal Block: Adductor Canal Block performed at mid-thigh level to block the saphenous nerve under guidance of a linear ultrasound transducer probe (General Electric; GE). Performed using a 22-gauge 2-inch Stimuplex A needle ( B. Braun Medical Inc., Melsungen, Germany).Solution to be injected will be a combination of Ropivacaine 0.2 % ( 0.5 ml/kg, maximum of 30 ml) and methylprednisolone acetate 1 mg/kg ( maximum of 40 mg ).
  .
Arm/Group | Adductor Canal Block | Femoral Nerve Block
Number analyzed (Participants) | 26 | 26
Kilogram-force (Kgf) | 1.1 [0.0 to 25.6] | 0.0 [0.0 to 15.3]
Statistical Analysis 1: Comparison: Adductor Canal Block vs Femoral Nerve Block; Test type: Other — Test of difference was conducted; p = 0.026, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Post-operative Pain Scores Using the Numeric Pain Scoring System (NS)
Description: Assessed by Numeric Scale (NS) pain scoring system. Minimum 0 and maximum 10 . Higher scores means worse outcome (pain)
Time Frame: 4 hours and 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Adductor Canal Block | Femoral Nerve Block
Number analyzed (Participants) | 26 | 26
score on a scale
  4 hours post block | 4.5 [2.0 to 5.0] | 4.5 [4.0 to 6.0]
  24 hours post block | 5.0 [3.0 to 7.0] | 6.0 [5.0 to 7.0]
Statistical Analysis 1: Comparison: Adductor Canal Block vs Femoral Nerve Block; Test type: Other; p = 0.762, Wilcoxon (Mann-Whitney) — Alpha = 0.025 for multiple comparisons
Statistical Analysis 2: Comparison: Adductor Canal Block vs Femoral Nerve Block; Test type: Other; p = 0.410, Wilcoxon Rank Sum Test with Exact Option — Alpha = 0.025 for multiple comparisons

3. Primary Outcome: Total Opioid Consumption at 24 Hours Post-block
Description: Total intravenous morphine/morphine equivalent consumption in milligrams (mg) at 24 hours post-block
Time Frame: 24 hours following peripheral nerve block performance.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Adductor Canal Block | Femoral Nerve Block
Number analyzed (Participants) | 26 | 26
milligrams | 28.9 (9.0) | 26.9 (9.4)
Statistical Analysis 1: Comparison: Adductor Canal Block vs Femoral Nerve Block; Test type: Other — Test of Difference conducted; p = 0.454, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Death, serious adverse events, and other adverse events were not assessed for participants in the study
Description: Death, serious adverse events, and other adverse events were not assessed for participants in the study
Arm/Group | Adductor Canal Block | Femoral Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The sample size analysis was known to be limited due to population differences between our site and the site referenced. Due to feasibility issues the study was concluded as planned with completed enrollment of 52 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT03053401/Prot_SAP_000.pdf